CLINICAL TRIAL: NCT00143403
Title: Multi-Centre Phase III Open Label Randomized Trial Comparing CPT-11 In Combination With A 5-FU/FA Infusional Regimen To The Same 5-FU/FA Infusional Regimen Alone, As Adjuvant Treatment After Resection Of Liver Metastases For Colorectal Cancer.
Brief Title: Comparing Irinotecan and 5 FU/FA To 5-FU/FA After Resection Of Liver Metastases For Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPT-GMA-301; A5961076
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Results first posted 2009-06-01 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Colorectal Neoplasms; Liver Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms; Liver Neoplasms | interventions — Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Irinotecan + 5 FU + folinic acid
- 2 (Active Comparator)
  Interventions: Drug: Folinic Acid + 5 FU

INTERVENTIONS:
Drug: Irinotecan + 5 FU + folinic acid — irinotecan 180 mg/m2 folinic acid 400 mg/m2 (DL) followed by 5 FU bolus 400 mg/m2 5 FU continuous infusion (2400 mg/m2 over 46 hours) every 2 weeks
  Arms: 1
Drug: Folinic Acid + 5 FU — folinic acid 400 mg/m2(DL) followed by bolus 5 FU 400mg/m2 5 FU continuous infusion (2400 mg/m2 over 46 hours) every 2 weeks
  Arms: 2

SUMMARY:
To see if Disease Free Survival (DFS) is improved when complete surgical resection of liver metastases (R0) is followed by chemotherapy with CPT-11 and 5-FU/FA as FOLFIRI regimen, compared to 5-FU/FA alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the colon or rectum with complete resection of primary tumour.
* Complete surgical resection (R0) of the liver metastasis(es) within a minimum of 3 weeks, and a maximum of 8 weeks prior to the first study treatment infusion.
* Exclusively hepatic metastasis (es) : absence of bone, lung and brain metastases.

Exclusion Criteria:

* Prior hepatic radiation or resection.
* Prior radiofrequency ablation or cryoablation Incomplete surgical resection of liver metastasis (es).
* Prior chemotherapy for metastatic disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2001-12; Primary Completion 2008-02 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (60):
- Belgium (2):
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Roeselare
- Denmark (3):
  - Pfizer Investigational Site, Copenhagen
  - Pfizer Investigational Site, Herlev
  - Pfizer Investigational Site, Odense
- France (13):
  - Pfizer Investigational Site, Amiens
  - Pfizer Investigational Site, Avignon
  - Pfizer Investigational Site, Boulogne-Billancourt
  - Pfizer Investigational Site, Clermont-Ferand Cedex 1
  - Pfizer Investigational Site, Colmar
  - Pfizer Investigational Site, Grenoble
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Nîmes
  - Pfizer Investigational Site, Rennes
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Toulouse
- Germany (10):
  - Pfizer Investigational Site, Cottbus
  - Pfizer Investigational Site, Dessau
  - Pfizer Investigational Site, Erlangen
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Magdeburg
  - Pfizer Investigational Site, Mainz
  - Pfizer Investigational Site, Oldenburg
  - Pfizer Investigational Site, Regensburg
  - Pfizer Investigational Site, Tübingen
- Pfizer Investigational Site, Hong Kong, Hong Kong
- Israel (5):
  - Pfizer Investigational Site, Haifa
  - Pfizer Investigational Site, Petah Tikva
  - Pfizer Investigational Site, Rehovot
  - Pfizer Investigational Site, Tel Aviv
  - Pfizer Investigational Site, Tel Litwinsky
- Italy (8):
  - Pfizer Investigational Site, Carpi, Modena
  - Pfizer Investigational Site, Brescia
  - Pfizer Investigational Site, Latisana, UD
  - Pfizer Investigational Site, Padua
  - Pfizer Investigational Site, Parma
  - Pfizer Investigational Site, Piacenza
  - Pfizer Investigational Site, Reggio Emilia
  - Pfizer Investigational Site, Rozzano (Mi)
- Pfizer Investigational Site, Porto, Portugal
- Pfizer Investigational Site, Panorama, Cape Town, South Africa
- South Korea (3):
  - Pfizer Investigational Site, Daegu
  - Pfizer Investigational Site, Goyang
  - Pfizer Investigational Site, Seoul
- Spain (5):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona
  - Pfizer Investigational Site, Santander, Cantabria
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Seville, Sevilla
- Pfizer Investigational Site, Gothenburg, Sweden
- Pfizer Investigational Site, Bern, Switzerland
- Pfizer Investigational Site, Taoyuan District, Taiwan
- Ukraine (2):
  - Pfizer Investigational Site, Donetsk, Ukraine
  - Pfizer Investigational Site, Kiev
- United Kingdom (3):
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Southampton
  - Pfizer Investigational Site, Surrey

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=CPT-GMA-301&StudyName=Comparing%20Irinotecan%20and%205%20FU/FA%20To%205-FU/FA%20After%20Resection%20Of%20Liver%20Metastases%20For%20Colorectal%20Cancer

RESULTS

PARTICIPANT FLOW:
Recruitment Details: study was conducted at 66 centers.
Pre-assignment Details: Eligible subjects (subjects who underwent complete liver metastasis resection within 8 weeks of study drug administration) were randomly assigned. Of the 321 subjects randomized in the study, all but 15 were treated.
Groups:
- 5-FU/FA: simplified 5-FU/FA De Gramont regimen for a period of twelve 2-week cycles (6 months)
- Irinotecan + 5-FU/FA: irinotecan plus simplified 5-FU/FA De Gramont regimen for a period of twelve 2-week cycles (6 months)
Period: Overall Study
Arm/Group | 5-FU/FA | Irinotecan + 5-FU/FA
Started | 160 | 161
Treated | 153 | 153
Completed | 125 (Received maximum number of cycles.) | 115 (Received maximum number of cycles.)
Not Completed | 35 | 46
Not completed — Adverse Event | 3 | 8
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 3 | 12
Not completed — Relapse | 15 | 7
Not completed — Protocol Violation | 2 | 2
Not completed — specified by site | 4 | 9
Not completed — Randomized Not Treated | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5-FU/FA | Irinotecan + 5-FU/FA | Total
Number analyzed (Participants) | 153 | 153 | 306
Age Continuous [Median (Full Range); unit: years] | 61 [34 to 76] | 63 [27 to 75] | 62 [27 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 63 | 116.0
  Male | 100 | 90 | 190.0

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival (DFS)
Description: time interval between the date of randomization and the earliest date of local, regional or distant relapse, or death due to cancer.
Time Frame: last tumor assessment date or cut-off date, whichever is earlier.
Population: Full analysis set = all treated subjects according to randomization: n=153, 153 for 5-FU/FA & Irinotecan + 5-FU/FA, respectively. Safety analysis set (for Adverse Events) = all treated subjects according to treatment actually received (1 subject randomized to 5-FU/FA actually received treatment from Irinotecan + 5-FU/FA). n=152, 154 as above).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 5-FU/FA | Irinotecan + 5-FU/FA
Number analyzed (Participants) | 153 | 153
months | 21.6 [14.6 to 30.4] | 24.7 [18.7 to 38.9]
Statistical Analysis 1: Comparison: 5-FU/FA vs Irinotecan + 5-FU/FA; Test type: Superiority or Other; Hazard Ratio (HR) = 0.90, 95% CI [0.67 to 1.20] — HR: Irinotecan+5-FU/FA / 5-FU/FA
Statistical Analysis 2: Comparison: 5-FU/FA vs Irinotecan + 5-FU/FA; Test type: Superiority or Other; p = 0.468, Log Rank

2. Secondary Outcome: Overall Survival Rates
Description: Probability of being alive was calculated in a yearly increment.
Time Frame: Median follow-up time (42 months)
Population: as for outcome 1
Measure: Number; unit: survival rate
Arm/Group | 5-FU/FA | Irinotecan + 5-FU/FA
Number analyzed (Participants) | 153 | 153
survival rate
  12 months | 0.961 | 0.973
  24 months | 0.845 | 0.881
  36 months | 0.716 | 0.727

ADVERSE EVENTS:
Arm/Group | 5-FU/FA | Irinotecan + 5-FU/FA
Serious Adverse Events (participants affected / at risk) | 15/152 | 32/154
Other Adverse Events (participants affected / at risk) | 146/152 | 150/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5-FU/FA (N=152) | Irinotecan + 5-FU/FA (N=154)
Abdominal pain NOS (Gastrointestinal disorders) | 2 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Anaemia NOS (Blood and lymphatic system disorders) | 0 | 1
Appendicitis (Gastrointestinal disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Axillary vein thrombosis (Vascular disorders) | 0 | 1
Cardiac disorder NOS (Cardiac disorders) | 0 | 1
Catheter related complication (General disorders) | 0 | 1
Catheter related infection (Infections and infestations) | 1 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Chest pain (General disorders) | 0 | 2
Cholecystitis acute NOS (Hepatobiliary disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Depression (Psychiatric disorders) | 0 | 1
Device failure (Injury, poisoning and procedural complications) | 1 | 0
Diarrhoea NOS (Gastrointestinal disorders) | 0 | 7
Dizziness (Nervous system disorders) | 0 | 3
Enteritis (Gastrointestinal disorders) | 1 | 0
Gait abnormal (General disorders) | 0 | 1
Hepatic disorder NOS (Hepatobiliary disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Injection site thrombosis (General disorders) | 0 | 1
Intestinal obstruction NOS (Gastrointestinal disorders) | 2 | 0
Liver abscess (Infections and infestations) | 0 | 2
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 3
Neutropenic sepsis (Infections and infestations) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Peripheral swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Phlebitis NOS (Vascular disorders) | 0 | 1
Pneumothorax NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 2
Rectovaginal fistula (Gastrointestinal disorders) | 0 | 1
Renal impairment NOS (Renal and urinary disorders) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Tachycardia NOS (Cardiac disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 1
Vomiting NOS (Gastrointestinal disorders) | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 5-FU/FA (N=152) | Irinotecan + 5-FU/FA (N=154)
Abdominal pain upper (Gastrointestinal disorders) | 17 | 22
Abdominal pain, NOS (Gastrointestinal disorders) | 40 | 41
Alopecia (Skin and subcutaneous tissue disorders) | 28 | 69
Anemia NOS (Blood and lymphatic system disorders) | 19 | 21
Anorexia (Metabolism and nutrition disorders) | 21 | 32
Anxiety (Psychiatric disorders) | 2 | 9
Appetite decreased NOS (Metabolism and nutrition disorders) | 8 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 10
Asthenia (General disorders) | 48 | 53
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 10
Cholinergic syndrome (Nervous system disorders) | 1 | 17
Conjunctivitis (Eye disorders) | 9 | 2
Constipation (Gastrointestinal disorders) | 30 | 46
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 13
Diarrhea, NOS (Gastrointestinal disorders) | 80 | 98
Dizziness (Nervous system disorders) | 14 | 12
Dysgeusia (Nervous system disorders) | 19 | 10
Dyspepsia (Gastrointestinal disorders) | 15 | 14
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 9 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 19
Fatigue (General disorders) | 28 | 34
Flatulence (Gastrointestinal disorders) | 3 | 8
Headache (Nervous system disorders) | 23 | 22
Insomnia (Psychiatric disorders) | 14 | 11
Lacrimation increased (Eye disorders) | 13 | 12
Leukopenia NOS (Blood and lymphatic system disorders) | 10 | 27
Mucosal inflammation NOS (General disorders) | 31 | 32
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 10 | 8
Nausea (Gastrointestinal disorders) | 91 | 116
Neutropenia (Blood and lymphatic system disorders) | 25 | 62
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 25 | 20
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Pigmentation disorder NOS (Skin and subcutaneous tissue disorders) | 13 | 7
Pyrexia (General disorders) | 10 | 13
Rhinitis NOS (Respiratory, thoracic and mediastinal disorders) | 11 | 9
Stomatitis (Gastrointestinal disorders) | 40 | 34
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 4
Vomiting, NOS (Gastrointestinal disorders) | 37 | 64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.